CLINICAL TRIAL: NCT07364721
Title: Comparative Efficacy of Maitland Mobilization vs. McKenzie Press-Up in Chronic Low Back Pain: A Randomized Trial
Brief Title: Maitland Mobilization vs. McKenzie Press-Up in Chronic LBP
Acronym: LBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palestine Ahliya University (Other)
Responsible Party: Principal Investigator, Azzam Alarab, Chairperson, Department of Medical Sciences - Master's, Palestine Ahliya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Palestine Ahliya U
Record Dates: First submitted 2026-01-03; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Back Pain Lower Back
Keywords: McKenzie Exercise; Low back pain; Posteroanterior mobilization
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: The treatment techniques applied to the two groups are as follows. Group A (Central PA Maitland mobilization with MFR): 25 patients received 3 sessions per week for 4 weeks; the central PA mobilization technique was applied for 10 minutes and MFR for 20 minutes (30 seconds break each five minutes). Group B (McKenzie PPU exercise with MFR): 25 patients received three sessions per week for four weeks, with each session consisting of 10 minutes of McKenzie PPU exercise followed by 20 minutes of MFR, also with a 30-second break every five minutes.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1- Group A :Central PA Maitland mobilization with MFR (Experimental): Central PA Maitland mobilization with MFR
  Interventions: Other: Group B (McKenzie PPU exercise with MFR); Other: McKenzie PPU exercise with MFR
- Arm 2- Group B:McKenzie PPU exercise with MFR (Experimental): Patient position: The patient assumes a prone position. investigator position: The investigator stands beside the patient and provides verbal instruction.
  Direction: Patients were being instructed to perform PPU exercise by using their upper limbs to push their upper body up into spinal extension while the pelvis remained on the treatment table. The patient is trained to extend the lumbar spine to the maximum pain-free range.
  Frequency: Ten repetitions for three sets with a 30-second break between each set for almost 10 minutes [27].
  Interventions: Other: Group B (McKenzie PPU exercise with MFR); Other: Central Posteroanterior Mobilization

INTERVENTIONS:
Other: Group B (McKenzie PPU exercise with MFR) — Patient position: The patient assumes a prone position. Therapist position: The therapist stands beside the patient and provides verbal instruction.
  Direction: Patients were being instructed to perform PPU exercise by using their upper limbs to push their upper body up into spinal extension while the pelvis remained on the treatment table. The patient is trained to extend the lumbar spine to the maximum pain-free range.
  Frequency: Ten repetitions for three sets with a 30-second break between each set for almost 10 minutes
Other: Central Posteroanterior Mobilization — According to Maitland's concept, mobilization technique including passive accessory intervertebral movement was applied to cause movement in the stiff vertebral segment without the active involvement of the muscles [44]. Central PA mobilization technique is a cornerstone of Maitland vertebral mobilization [38]. It can be achieved by passive force onto a vertebral segment in the PA direction [44].
  Patient position: When applying this technique, the patient assumes a relaxed and comfortable prone position, with the arms positioned alongside the body [23, 24].
  investigator position: The investigator stands close to the patient, with their sternum perpendicular to the selected lumbar spinous process [23]. The investigator uses the ulnar surface of the hand (pisiform) over the selected spinous process in the lumbar spine, another hand taken was placed above the first hand to reinforce, and the elbow should slightly bent with forearm in neutral between supination & pronation.
  Arms: Arm 2- Group B:McKenzie PPU exercise with MFR
Other: McKenzie PPU exercise with MFR — Patient position: The patient assumes a prone position. investigator position: The investigator stands beside the patient and provides verbal instruction.
  Direction: Patients were being instructed to perform PPU exercise by using their upper limbs to push their upper body up into spinal extension while the pelvis remained on the treatment table. The patient is trained to extend the lumbar spine to the maximum pain-free range.
  Frequency: Ten repetitions for three sets with a 30-second break between each set for almost 10 minutes
  Arms: Arm 1- Group A :Central PA Maitland mobilization with MFR

SUMMARY:
ABSTRACT Objective:This study aimed to compare the efficacy of central posteroanterior (PA) Maitland mobilization with myofascial release (MFR) and McKenzie prone press-up (PPU) exercise with MFR in the treatment of adult patients with chronic non-specific low back pain (CNLBP). Materials and Methods:A randomized controlled trial was conducted at Salhab Center and Al Shifa's Specialized Complex in Bethlehem between January 2023 and May 2024. The study included 50 adult patients (aged 18-50) with CNLBP of more than 3 months but less than 2 years' duration, referred by an orthopedic specialist at Beit Sahour Medical Center. Participants were randomly assigned to two groups: one received central PA Maitland mobilization with MFR, and the other received McKenzie PPU exercise with MFR. Pain intensity, functional impairment, and fear-avoidance beliefs were assessed using the Visual Analog Scale (VAS), Oswestry Disability Index (ODI), and Fear-Avoidance Beliefs Questionnaire (FABQ). Each patient underwent three sessions per week for four weeks.

DETAILED DESCRIPTION:
This randomized controlled trial evaluated physiotherapy interventions in adults with chronic non-specific low back pain (CNLBP). The study was conducted at Salhab Center for Physiotherapy and Al Shifa's Specialized Complex in Bethlehem City between December 2023 and May 2024. These centers were selected for their accessibility and coordinated referral system.

Participants were referred from orthopedic assessment to physiotherapy, where baseline evaluations were completed prior to randomization. Random allocation to intervention groups was performed using a concealed allocation method.

Physiotherapy interventions were delivered by licensed physiotherapists according to standardized treatment protocols to ensure consistency. Treatment sessions consisted of structured therapeutic exercises and manual therapy techniques, with progression individualized based on patient response. Outcome data were collected at baseline and at the end of the intervention period using validated assessment tools. Participant adherence and adverse events were monitored throughout the study. All procedures were conducted in accordance with ethical standards, and informed consent was obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

* 18 and 50 years of age,
* Male or female, with NSLBP localized between the lower rib and the gluteal fold
* Persisting for more than three months and occurring on at least half of the days in the past three months, with pain affecting daily functional activities.
* VAS score between 40 mm and 80 mm at the initial assessment
* No use of NSAID medications during treatment sessions.

Exclusion Criteria:

* Patients younger than 18 or older than 50 years,
* Those with mental health disorders, systemic or neurological diseases, or specific spinal pathologies such as facet joint dysfunction, piriformis syndrome, disc herniation, spinal tumors, spondylitis, spondylolisthesis, spinal stenosis, or spinal osteoporosis. Patients were also excluded if they had contraindications to mobilization, a history of spinal surgery or epidural injections, physiotherapy for LBP within the last six months, a VAS score outside the 40-80 mm range, pregnancy, or a current upper limb injury.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index | 4 WEEKS
  0% (no disability) to 100% (severe disability)

OTHER OUTCOMES:
Visual Analogu Scale | 4 WEEKS
  0 no pain , 10 severe pain
Fear-Avoidance Belief Questionnaire | 4 WEEKS
  The Fear Avoidance Beliefs Questionnaire (FABQ) scoring involves summing responses to 16 items on a 0-6 Likert scale (0=completely disagree, 6=completely agree

CONTACTS AND LOCATIONS:
Locations (1):
- Palestine Ahliya University, Bethlehem, West Bank, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No